CLINICAL TRIAL: NCT04708535
Title: Adaptive Immune Response in Visceral and Subcutaneous Fat: Role in Human Insulin Resistance
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Principal Investigator, Stanford University
Other Study IDs: 40196; 1-19-ICTS-073 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2018-07-03; First posted 2021-01-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Insulin Resistance; Insulin Sensitivity; Obesity; Inflammation
MeSH Terms: conditions — Insulin Resistance; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Visceral adipose tissue (VAT), Subcutaneous adipose tissue (SAT) and peripheral blood samples are obtained perioperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric Cohort: For consenting subjects who are undergoing bariatric surgery, a visceral fat sample will be taken during surgery. In addition to the fat sample, insulin resistance will be measured and determined by a modification of the insulin suppression test.

SUMMARY:
The proposed study is designed to test the hypothesis that in human obesity, the balance of pro- and anti-inflammatory T cells in fat tissue is in fact related to macrophage phenotype and insulin resistance, and how it is related.

This study is needed to confirm whether conclusions based on studies of visceral adipose tissue in mice are indeed applicable to humans.

We also want to determine the relationship between insulin resistance/hyperinsulinemia and ability to lose weight in obese individuals.

DETAILED DESCRIPTION:
Previous studies have found convincing evidence of the relationship between insulin resistance, T cell profiles, macrophage profiles and inflammation of the fat cells. This study will add human subjects to that body of evidence.

Overview Aim 1: Test the hypothesis that the balance of anti- inflammatory vs proinflammatory T cells is protective for systemic insulin resistance. T cell profiles in subcutaneous and visceral tissue and blood will be compared in IR vs IS obese humans at baseline and potentially after 12 months following weight loss. Tcell profile will be evaluated for relationships with IR and inflammation, with adjustment for total body fat. Secondarily, they will be evaluated for relationship to adipose cell size.

Overview Aim 2: Test the hypothesis that macrophage phenotype in adipose tissue is associated with T cell profile and IR. Frequency of macrophage phenotypes (M1 vs M2) will be analyzed in IR vs IS obese humans at baseline and potentially after 12 months following weight loss.

Overview Aim 3: Testing the hypothesis insulin resistance is associated with T cell receptor phenotypes in subcutaneous and visceral tissue. IR and IS subjects will be evaluated at baseline by sequencing of expressed TCRs in paired SAT, VAT, and blood. We will determine whether TCR phenotypes are shared between different IR individuals.

ELIGIBILITY:
Inclusion Criteria:

* Current patients of Stanford Healthcare, Bariatric Surgery Clinic, scheduled to undergo bariatric surgery (sleeve or RYGB)
* BMI 30-55kg/m2
* 30-65 years of age
* good general health, no major organ disease
* non-diabetic by current American Diabetes Association (ADA) criteria (fasting glucose <126mg/dl)

Exclusion Criteria:

* Subjects with any clinical or biochemical evidence of significant anemia, gastrointestinal, cardiac, hepatic or renal disease will be excluded.
* Subjects with other medical problems may participate as long as the problems are stable.
* Subjects with active psychiatric disorders or past history of bariatric surgery
* Pregnant or lactating women will also be excluded from the study, due to possible risk to the fetus or infant.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are no restrictions in regards to gender, race, or socioeconomic status. The racial/ ethnic composition of the study population will be reflective of the communities surrounding the Stanford University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
T-cell profile in visceral and subcutaneous fat | baseline (within 2 months prior to bariatric surgery)
  Pro-inflammatory and anti-inflammatory T cell profiles in subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.
T-cell profile in visceral and subcutaneous fat | post-operatively (1-2 years status post bariatric surgery)
  Pro-inflammatory and anti-inflammatory T cell profiles in subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.
Adipose cell size associated with T cell profile and IR. | baseline (within 2 months prior to bariatric surgery)
  Cell size of subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.
Adipose cell size associated with T cell profile and IR. | post-operatively (1-2 years status post bariatric surgery)
  Cell size of subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.
Macrophage phenotype | (Timeframe: baseline (within 2 months prior to bariatric surgery)
  Frequency of macrophage phenotype (M1 vs M2) in subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.
Macrophage phenotype | post-operatively (1-2 years status post bariatric surgery)
  Frequency of macrophage phenotype (M1 vs M2) in subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.
T cell receptor phenotypes | (Timeframe: baseline (within 2 months prior to bariatric surgery)
  Frequency of T-cell receptors in subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.
T cell receptor phenotypes | post-operatively (1-2 years status post bariatric surgery)
  Frequency of T-cell receptors in subcutaneous adipose tissue and visceral adipose tissue measured via flow cytometry.

SECONDARY OUTCOMES:
Change in body weight | (Timeframe: baseline (within 2 months prior to bariatric surgery)
  Percent body weight loss post bariatric surgery, accounting for insulin sensitivity, T-cell profile, cell size, and macrophage and T-cell phenotypes.
Change in body weight | post-operatively (1-2 years status post bariatric surgery)
  Percent body weight loss post bariatric surgery, accounting for insulin sensitivity, T-cell profile, cell size, and macrophage and T-cell phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No